CLINICAL TRIAL: NCT02447250
Title: Albuterol Dose-Response on Pulmonary Function Testing in Preterm Infants at Risk of Bronchopulmonary Dysplasia
Brief Title: Preterm Infant Inhaled Albuterol Dosing
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Cynthia McEvoy, Associate Professor of Pediatrics, Oregon Health and Science University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB00009883
Record Dates: First submitted 2015-05-14; First posted 2015-05-18 (Estimated); Results first posted 2019-05-23 (Actual); Last update posted 2019-05-23 (Actual); Status verified 2019-05

CONDITIONS: Bronchopulmonary Dysplasia; Very Low Birth Weight
Keywords: Bronchopulmonary dysplasia; very low birth weight; albuterol; pulmonary function test
MeSH Terms: conditions — Bronchopulmonary Dysplasia | interventions — Albuterol; Procaterol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single Arm: varied albuterol dose response (Experimental): Subjects will be evaluated in 3 sessions. The sessions will occur within a 7 day time span, beginning after 14 days of age and at 28w0d to 33w6d corrected gestational age. In each session, pulmonary function tests (PFTs) will be performed prior to and 15 minutes after a dose of albuterol. The dose will be different in each session. In the first session, a single dose of 180 micrograms (2 puffs) of albuterol sulfate via metered dose inhaler. The dose will be 270 micrograms in the second session and 360 micrograms in the third session. PFTs will be performed during quiet sleep while the baby is spontaneously breathing or while the baby is intubated and receiving mechanical ventilation. Resistance and compliance will be measured using the single breath occlusion technique.
  Interventions: Drug: Varied albuterol dose response

INTERVENTIONS:
Drug: Varied albuterol dose response — Subjects will be evaluated in 3 sessions. The sessions will occur within a 7 day time span, beginning between 14 or more days from birth and at a corrected gestational age of 28w0d to 33w6d. In each session, pulmonary function tests (PFTs) will be performed prior to and 15 minutes after a dose of albuterol. The dose will be different in each session. In the first session, a sinlge dose of 180 micrograms (2 puffs) of albuterol sulfate via metered dose inhaler. The dose will be 270 micrograms in the second session and 360 micrograms in the third session. PFTs will be performed during quiet sleep while the baby is spontaneously breathing or while the baby is intubated and receiving mechanical ventilation. Resistance and compliance will be measured using the single breath occlusion technique.
  Other Names: Albuterol sulfate; Salbutamol; Proventil; ProAir; Ventolin

SUMMARY:
The purpose of this study is to help determine the best dose of inhaled albuterol sulfate in premature babies at risk of developing bronchopulmonary dysplasia (BPD). BPD is the chronic lung disease of prematurity and is associated with increased morbidity and mortality, longer hospital stays, and increased healthcare utilization. Albuterol is an inhaled medication frequently used in premature infants with chronic lung disease and in people with asthma. It is believed to be safe, but the optimal dose for infants is not clear. The investigators hypothesize that albuterol may help a subset of premature infants with lung disease, but they need to determine the best dose prior to doing research about how effective it is for chronic lung disease/BPD. Response to each of three doses of albuterol will be measure using pulmonary function tests.

DETAILED DESCRIPTION:
1. Recruitment: Subjects at risk for developing bronchopulmonary dysplasia will be recruited from the Doernbecher Neonatal Care Center (DNCC).The subjects' mother will be approached by the investigators and consent obtained if she agrees to participate.
2. Medical Record and Interview: Information about the pregnancy, delivery, and neonatal course will be obtained from the medical record. This will include maternal body mass index (BMI) at first prenatal visit, maternal age and parity, birthweight, gestational age at birth, history of maternal betamethasone for fetal lung maturation, indication for preterm delivery (e.g. pre-eclampsia, preterm labor), surfactant administration, history of intubations and duration of mechanical ventilation in the infant, current level of respiratory support, use of diuretics, bronchodilators, and corticosteroids in the neonate. A brief interview will also be obtained from the subject's mother. The questions asked will involve tobacco exposure during the pregnancy and family history of asthma. The purpose of the data collected on the infant's mother is to help identify factors that may predict which premature infants will respond to albuterol.
3. Procedures: Pulmonary function tests (PFTs) are the procedures involved in this study. PFTs are non-invasive, require no sedation, and are commonly used to provide standard medical care to preterm infants in the DNCC. PFTs involve placing a mask over the nose and mouth during quiet sleep. We will record flow-volume loops with passive respiration and measure respiratory compliance and passive respiratory resistance (Rr) using the single breath occlusion technique. A dose of albuterol will be given after baseline measurements are obtained; the PFTs will be repeated 15 minutes after administration. The testing will be the same for each of the three sessions, except the dose of albuterol will be altered each session (see below). There will be only one session per day, and all three sessions will occur within a 7 day period. Vital signs (respiratory rate, heart rate, oxygen saturation) will be continuously monitored during the testing.
4. Study Drug: Albuterol is a bronchodilator frequently prescribed in neonatal ICUs to help treat the symptoms of BPD. About 50% of preterm infants in the DNCC with evolving BPD have shown an improvement in their PFT after 2 puffs (180 micrograms) of albuterol (unpublished data). The typical dosing is 2-4 puffs every 4-6 hours but the optimal dose in premature infants is not known. In this study, 2 puffs (180 micrograms) will be given on the first day of PFTs, 3 puffs (270 micrograms) the second day, and 4 puffs (260 micrograms) on the third day.

ELIGIBILITY:
Inclusion Criteria:

* very low birthweight infant (<1500g)
* gestational age at birth <32 weeks
* age 14 or more days and corrected to 28w0d to 33w6d gestational age
* continuing to require respiratory support and/or supplemental oxygen

Exclusion Criteria:

* chromosomal abnormalities
* major congenital anomalies
* congenital heart disease, except atrial septal defect and patent ductus arteriosus
* clinical providers determine subject too unstable to undergo pulmonary function testing

Min Age: 14 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2013-10-24 (Actual); Primary Completion 2014-12-30 (Actual); Study Completion 2014-12-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia McEvoy, MD, MCR, Principal Investigator — Oregon Health and Science University; Amanda Kim, MD, Study Director — Oregon Health and Science University
Locations (1):
- Doernbecher Neonatal Care Center at Oregon Health & Science University, Portland, Oregon, United States

REFERENCES:
- [Background] Blake K, Madabushi R, Derendorf H, Lima J. Population pharmacodynamic model of bronchodilator response to inhaled albuterol in children and adults with asthma. Chest. 2008 Nov;134(5):981-989. doi: 10.1378/chest.07-2991. Epub 2008 Jun 26. PMID 18583517
- [Background] Ng G, da Silva O, Ohlsson A. Bronchodilators for the prevention and treatment of chronic lung disease in preterm infants. Cochrane Database Syst Rev. 2012 Jun 13;(6):CD003214. doi: 10.1002/14651858.CD003214.pub2. PMID 22696334
- [Background] Jobe AH, Bancalari E. Bronchopulmonary dysplasia. Am J Respir Crit Care Med. 2001 Jun;163(7):1723-9. doi: 10.1164/ajrccm.163.7.2011060. No abstract available. PMID 11401896

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 1 subject was consented into the study, but then became too clinically unstable to participate in the study and remained unstable throughout the eligibility period.
Groups:
- Single Arm: Varied Albuterol Dose Response: Subjects will be evaluated in three sessions within a 7 day time span, beginning after 14 days of age and at 28w0d to 33w6d corrected gestational age. In each session, pulmonary function tests (PFTs) will be performed prior to and 15 minutes after a dose of albuterol. The dose will be different in each session. In the first session, a single dose of 180 micrograms (2 puffs) of albuterol sulfate via metered dose inhaler. The dose will be 270 micrograms in the second session and 360 micrograms in the third session. PFTs will be performed during quiet sleep while the baby is spontaneously breathing or while the baby is intubated and receiving mechanical ventilation. Resistance and compliance will be measured using the single breath occlusion technique.
  Varied albuterol dose response: Subjects will be evaluated in three sessions. The sessions will occur within a 7 day time span, beginning between 14 or more days from birth and at a corrected gestational age of 2
Period: First Dose (180 mcg Albuterol)
Arm/Group | Single Arm: Varied Albuterol Dose Response
Started | 14
Completed | 14
Not Completed | 0
Period: Second Dose (270 mcg Albuterol)
Arm/Group | Single Arm: Varied Albuterol Dose Response
Started | 14
Completed | 13
Not Completed | 1
Not completed — elevated HR with first dose | 1
Period: Third Dose (360 mcg Albuterol)
Arm/Group | Single Arm: Varied Albuterol Dose Response
Started | 13
Completed | 8
Not Completed | 5
Not completed — Clinically unstable, unable to do PFT | 1
Not completed — Elevated HR with 2nd dose | 4

BASELINE CHARACTERISTICS:
Arm/Group | Single Arm: Varied Albuterol Dose Response
Number analyzed (Participants) | 14
Age, Continuous [Mean (Full Range); unit: days] | 36 [17 to 66]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 4
birthweight [Mean (Full Range); unit: grams] | 895 [350 to 1293]
gestational age at birth [Mean (Full Range); unit: weeks] | 26.9 [24.1 to 29.9]
respiratory support at study entry, CPAP [Count of Participants; unit: Participants] | 12
respiratory support at study entry, mechanical ventilation [Count of Participants; unit: Participants] | 2
history of any mechanical ventilation [Count of Participants; unit: Participants] | 8
received surfactant [Count of Participants; unit: Participants] | 7
received antenatal corticosteroids [Count of Participants; unit: Participants] | 13
ever received albuterol prior to study entry [Count of Participants; unit: Participants] | 0
received diuretics prior to study entry [Count of Participants; unit: Participants] | 3
reason for preterm delivery: preterm labor [Count of Participants; unit: Participants] | 6
maternal age, years (mean) [Mean (Full Range); unit: years] | 26.4 [17 to 36]
maternal BMI (mean, range) [Median (Full Range); unit: kg/ m^2] | 25.5 [18.7 to 47]
maternal diabetes mellitus (pregestational or gestational) [Count of Participants; unit: Participants] | 4
family history of asthma [Count of Participants; unit: Participants] | 2
maternal smoking during pregnancy [Count of Participants; unit: Participants] | 4
second hand smoke exposure during pregnancy [Count of Participants; unit: Participants] | 6

OUTCOME MEASURES:

1. Primary Outcome: Change in Respiratory Resistance
Description: The primary outcome is the percentage of subjects who show a positive response to each dose of albuterol. A positive response is defined as a greater than or equal to 10% decrease in respiratory resistance (Rrs). The change in RRs was measured at baseline and again after each dose of albuterol. All measurements were taken within a 7 day time frame for each subject such that each subject would have up to 3 results measured during a 7 day period, if he/she were able to complete three sets of PFTs according to study protocol. The change in Rrs was calculated by subtracting the baseline Rrs from the post-albuterol Rrs.
Time Frame: Within one week of performing pulmonary function tests
Population: Some subjects did not receive all 3 doses (based on how they tolerated initial dose(s))
Measure: Mean (Standard Deviation); unit: cm h2o/mL/sec
Groups:
- Single Arm: Varied Albuterol Dose Response: Subjects will be evaluated in 3 sessions. The sessions will occur within a 7 day time span, beginning after 14 days of age and at 28w0d to 33w6d corrected gestational age. In each session, pulmonary function tests (PFTs) will be performed prior to and 15 minutes after a dose of albuterol. The dose will be different in each session. In the first session, a single dose of 180 micrograms (2 puffs) of albuterol sulfate via metered dose inhaler. The dose will be 270 micrograms in the second session and 360 micrograms in the third session. PFTs will be performed during quiet sleep while the baby is spontaneously breathing or while the baby is intubated and receiving mechanical ventilation. Resistance and compliance will be measured using the single breath occlusion technique.
  Varied albuterol dose response: Subjects will be evaluated in three sessions. The sessions will occur within a 7 day time span, beginning between 14 or more days from birth and at a corrected gestational age of 2
Arm/Group | Single Arm: Varied Albuterol Dose Response
Number analyzed (Participants) | 11
cm h2o/mL/sec
  dose 1 | 0.011 (0.016)
  dose 2: number analyzed (Participants) | 10
  dose 2 | 0.006 (0.008)
  dose 3: number analyzed (Participants) | 6
  dose 3 | 0.014 (0.014)

2. Secondary Outcome: Number of Participants With Positive Response at Different Albuterol Doses
Description: Compare number of subjects who have a positive response (greater than or equal to 10% decrease in respiratory resistance) to each dose of albuterol
Time Frame: Data collected 15 minutes after dose in each session. Study includes 3 sessions within a 7 day period.
Population: Measuring Rrs can be technically challenging, particularly in premature infants, and we did not have measurable Rrs for every subject at every time point, therefore the denominator here is not the same as the total number of participants. For example, we have missing/unmeasurable Rrs for 3 subjects at the lowest albuterol dose.
Measure: Number; unit: participants
Groups:
- Single Arm: Varied Albuterol Dose Response: Subjects will be evaluated in 3 sessions. The sessions will occur within a 7 day time span, beginning after 14 days of age and at 28w0d to 33w6d corrected gestational age. In each session, pulmonary function tests (PFTs) will be performed prior to and 15 minutes after a dose of albuterol. The dose will be different in each session. In the first session, a single dose of 180 micrograms (2 puffs) of albuterol sulfate via metered dose inhaler. The dose will be 270 micrograms in the second session and 360 micrograms in the third session. PFTs will be performed during quiet sleep while the baby is spontaneously breathing or while the baby is intubated and receiving mechanical ventilation. Resistance and compliance will be measured using the single breath occlusion technique.
  Varied albuterol dose response: Subjects will be evaluated in 3 sessions. The sessions will occur within a 7 day time span, beginning between 14 or more days from birth and at a corrected gestational age of 28w0d to
Arm/Group | Single Arm: Varied Albuterol Dose Response
Number analyzed (Participants) | 14
participants
  positive Rrs response at 180 mcg albuterol: number analyzed (Participants) | 11
  positive Rrs response at 180 mcg albuterol | 6
  positive Rrs response at 270 mcg albuterol: number analyzed (Participants) | 10
  positive Rrs response at 270 mcg albuterol | 4
  positive Rrs response at 360 mcg albuterol: number analyzed (Participants) | 6
  positive Rrs response at 360 mcg albuterol | 4

3. Secondary Outcome: Birth Weight of Albuterol Responders vs Non Responders
Description: birth weight in grams of each subject was recorded at time of enrollment
Time Frame: within one week of entering study
Population: This data included 10 subjects who responded to albuterol at at least one dose, and 3 subjects who did not show a positive response to albuterol at any dose
Measure: Mean (Standard Deviation); unit: grams
Arm/Group | Single Arm: Varied Albuterol Dose Response
Number analyzed (Participants) | 13
grams
  albuterol responders: number analyzed (Participants) | 10
  albuterol responders | 847.2 (296)
  albuterol non responders: number analyzed (Participants) | 3
  albuterol non responders | 1147.7 (216)
Statistical Analysis 1: Comparison: Single Arm: Varied Albuterol Dose Response; comparison of mean birth weights between responders and non-responders; Test type: Other; p = 0.14, Chi-squared

4. Secondary Outcome: Gestational Age at Birth
Description: Average gestational age (GA) in weeks at birth for subjects who responded to albuterol versus subjects without a positive response
Time Frame: within one week of entering study
Population: We have data for 10 subjects who responded to albuterol and 3 subjects who did not respond.
Measure: Mean (Standard Deviation); unit: weeks
Arm/Group | Single Arm: Varied Albuterol Dose Response
Number analyzed (Participants) | 13
weeks
  birth GA albuterol responders, weeks: number analyzed (Participants) | 10
  birth GA albuterol responders, weeks | 26.7 (1.9)
  birth GA albuterol non responders: number analyzed (Participants) | 3
  birth GA albuterol non responders | 28.5 (1.2)
Statistical Analysis 1: Comparison: Single Arm: Varied Albuterol Dose Response; Test type: Other; p = 0.16, Chi-squared

5. Secondary Outcome: Etiology of Preterm Delivery
Description: Reason for each subject's preterm delivery was classified as either preterm labor or delivery for maternal indications (eg pre-eclampsia).
Time Frame: within one week of entering study
Population: 5 subjects were delivered due to preterm labor, and 8 delivered prematurely due to maternal indications
Measure: Count of Participants; unit: Participants
Arm/Group | Single Arm: Varied Albuterol Dose Response
Number analyzed (Participants) | 13
Participants
  preterm labor, responsive to albuterol: number analyzed (Participants) | 5
  preterm labor, responsive to albuterol | 4
  maternal indicated delivery, responsive to albuter: number analyzed (Participants) | 8
  maternal indicated delivery, responsive to albuter | 6
Statistical Analysis 1: Comparison: Single Arm: Varied Albuterol Dose Response; Test type: Other; p = 1.0, Fisher Exact

6. Other Pre Specified Outcome: Family History of Asthma and Likelihood to Respond to Albuterol
Description: Family history was obtained from verbal history by subject's mother at time of enrollment in study. A positive family history was noted if a first degree relative of the subject (infant) had a diagnosis of asthma.
Time Frame: History collected at enrollment, albuterol response assessed within one week
Population: only 2 subjects had a history of a first-degree relative (parent or sibling) with asthma
Measure: Number; unit: participants
Arm/Group | Single Arm: Varied Albuterol Dose Response
Number analyzed (Participants) | 14
participants
  family hx of asthma, respond to albuterol: number analyzed (Participants) | 2
  family hx of asthma, respond to albuterol | 1
  no fam hx asthma, respond to albuterol: number analyzed (Participants) | 12
  no fam hx asthma, respond to albuterol | 9

7. Other Pre Specified Outcome: Maternal BMI at Time of Pregnancy and Likelihood of Positive Response to Albuterol
Description: Maternal BMI will be obtained from her medial record, and she will be asked about weight gain during pregnancy at time of enrollment. Results will be compared for infants born to women with a normal BMI vs. those with obese BMI (>30).
Time Frame: Maternal information collected at enrollment; albuterol response assessed within one week
Population: We have BMI data on 13 mothers.
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | Single Arm: Varied Albuterol Dose Response
Number analyzed (Participants) | 13
kg/m^2
  mean BMI mothers of albuterol-responders , any dos: number analyzed (Participants) | 10
  mean BMI mothers of albuterol-responders , any dos | 27.4 (8.6)
  mean BMI mothers of albuterol non-responders: number analyzed (Participants) | 3
  mean BMI mothers of albuterol non-responders | 27.3 (3.5)
Statistical Analysis 1: Comparison: Single Arm: Varied Albuterol Dose Response; Test type: Other; p = 1.0, Chi-squared

8. Other Pre Specified Outcome: Association of Smoke Exposure During Pregnancy and Neonatal Response to Albuterol
Description: Mothers who smoked cigarettes during pregnancy and the rate of albuterol response of their infants
Time Frame: Smoking and second hand smoke exposure history will be obtained at enrollment. Albuterol response will be obtained within one week.
Population: We have data for 9 subjects whose mothers did not smoke and 4 subjects whose mothers smoked
Measure: Number; unit: participants
Arm/Group | Single Arm: Varied Albuterol Dose Response
Number analyzed (Participants) | 13
participants
  albuterol responders of mothers who smoked: number analyzed (Participants) | 4
  albuterol responders of mothers who smoked | 4
  albuterol responders of non-smoker mothers %: number analyzed (Participants) | 9
  albuterol responders of non-smoker mothers % | 6
Statistical Analysis 1: Comparison: Single Arm: Varied Albuterol Dose Response; Test type: Other; p = 0.50, Fisher Exact

ADVERSE EVENTS:
Groups:
- Single Arm: Varied Albuterol Dose Response: Subjects will be evaluated in 3 sessions. The sessions will occur within a 7 day time span, beginning after 14 days of age and at 28w0d to 33w6d corrected gestational age. In each session, pulmonary function tests (PFTs) will be performed prior to and 15 minutes after a dose of albuterol. The dose will be different in each session. In the first session, a single dose of 180 micrograms (2 puffs) of albuterol sulfate via metered dose inhaler. The dose will be 270 micrograms in the second session and 360 micrograms in the third session. Resistance and compliance will be measured using the single breath occlusion technique.
  Varied albuterol dose response: Subjects will be evaluated in 3 sessions. The sessions will occur within a 7 day time span, beginning between 14 or more days from birth and at a corrected gestational age of 28w0d to
Arm/Group | Single Arm: Varied Albuterol Dose Response
All-Cause Mortality (participants affected / at risk) | 0/14
Serious Adverse Events (participants affected / at risk) | 0/14
Other Adverse Events (participants affected / at risk) | 1/14
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single Arm: Varied Albuterol Dose Response (N=14)
elevated heart rate above predefined criteria (Cardiac disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No